CLINICAL TRIAL: NCT06412081
Title: The Value of Point-of-care Lung Ultrasound for Physiotherapy in Hospitalized Patients With Acute Respiratory Symptoms
Brief Title: Lung Ultrasound for Physiotherapy in Hospitalized Patients With Respiratory Complications
Status: Recruiting | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, William Poncin, PT, PhD, PhD, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Other Study IDs: LUS-physio
Record Dates: First submitted 2024-05-08; First posted 2024-05-14 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Respiratory Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the relevance of using point-of-care lung ultrasound (LUS) in modifying the physiotherapist's treatment plan for patients hospitalized in a general ward.

DETAILED DESCRIPTION:
Hospitalized patients often confront respiratory issues stemming from diverse causes, such as pneumonia. Physiotherapists rely on a range of clinical and imaging data to inform their treatment decisions. Yet, they face challenges due to the absence of readily accessible, sensitive, specific, and reliable measurements to tailor the most effective physical therapeutic interventions based on individual clinical scenarios. Point-of-care Lung Ultrasound (LUS) holds promise in addressing these existing gaps.

This study aims to evaluate the impact of integrating LUS into clinical practice by comparing physiotherapists' initial clinical assessments and treatment plans with those made after incorporating LUS findings in patients admitted to a general ward.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization in a general ward
* Acute respiratory symptoms (< 48h)
* Chest X-ray available within 24h before or after the use of LUS

Exclusion Criteria:

* Any conditions precluding the use of LUS (thoracic skin lesions, thoracic bandage, subcutaneous emphysema)
* Inability to understand instructions due to cognitive impairment or due to language barrier

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Hospitalization in a general ward in the University Hospital Saint-Luc.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of change of treatment plan | Before and Immediately after the use of LUS (10-min interval)
  Relative change of treatment plan after the results of LUS in relation to the total number of events

SECONDARY OUTCOMES:
Agreement between the events observed on LUS and the events observed on Chest X-Ray | At baseline
  Number of concordant findings between LUS and Chest X-Ray. Each pair of tests will be rated as "positive" (same findings are observed between LUS and Chest X-Ray) or "negative" (findings are different).

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium